CLINICAL TRIAL: NCT03042065
Title: Salbutamol in the Pediatric Emergencies: Nebulization Estimated Via AerogeN or Jet
Acronym: SIBILANT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2016-A01276-45
Record Dates: First submitted 2017-01-25; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Asthma
Keywords: pediatrics; asthma; nebulization; vibrating mesh; salbutamol; Efficiency
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vibrating Mesh nebulizer (Experimental): Receive in the same aerosol solution 5 mg of Salbutamol (Ventolin, Glaxo, 5 mg / ml solution for nebulization) mixed with 0.5 mg Ipratropium Bromide (0.25 mg / ml) by nebulization every 20 min For 3 doses during the first hour of treatment, using vibrating Mesh nebulizer
  Interventions: Device: vibrating Mesh nebulizer
- jet nebulizer (Active Comparator): Receive, in the same aerosol solution, 5 mg of Salbutamol (Ventolin, Glaxo, 5 mg / ml solution for nebulization) mixed with 0.5 mg Ipratropium Bromide (0.25 mg / ml) by nebulization every 20 min For 3 doses during the first hour of treatment, using a jet nebulizer
  Interventions: Device: jet nebulizer

INTERVENTIONS:
Device: vibrating Mesh nebulizer — Receive in the same aerosol solution 5 mg of Salbutamol (Ventolin, Glaxo, 5 mg / ml solution for nebulization) mixed with 0.5 mg Ipratropium Bromide (0.25 mg / ml) by nebulization every 20 min For 3 doses during the first hour of treatment, using vibrating Mesh nebulizer
  Arms: vibrating Mesh nebulizer
Device: jet nebulizer — Receive in the same aerosol solution 5 mg of Salbutamol (Ventolin, Glaxo, 5 mg / ml solution for nebulization) mixed with 0.5 mg Ipratropium Bromide (0.25 mg / ml) by nebulization every 20 min For 3 doses during the first hour of treatment, using jet nebulizer
  Arms: jet nebulizer

SUMMARY:
Controlled trial of nebulized salbutamol using jet nebulizer or vibrating mesh technology in children presenting with acute moderate to severe asthma.

DETAILED DESCRIPTION:
Asthma is a chronic (long-term) lung disease that inflames and narrows the airways. Asthma causes recurring periods of wheezing (a whistling sound when you breathe), chest tightness, shortness of breath, and coughing. The coughing often occurs at night or early in the morning. Sometimes asthma symptoms are mild and go away on their own or after minimal treatment with asthma medicine. Other times, symptoms continue to get worse. When symptoms get more intense and/or more symptoms occur, it is called an asthma attack. Asthma attacks also are called flare-ups or exacerbation.

International Study of Asthma and Allergies in Childhood (ISAAC) found that about 14% of the world's children were likely to have had asthmatic symptoms in the last year and, crucially, the prevalence of childhood asthma varies widely between countries, and between centers within countries studied. These conclusions resulted from ISAAC's groundbreaking survey of a representative sample of 798,685 children aged 13-14 years in 233 centers in 97 countries. (ISAAC also studied a younger age group of children (6-7 years) and the findings were generally similar to the older children). These adolescents were asked whether they had experienced wheeze in the preceding 12 months. Prevalence of recent wheeze varied widely. The highest prevalence (>20%) was generally observed in Latin America and in English-speaking countries of Australasia, Europe and North America as well as South Africa. The lowest prevalence (<5%) was observed in the Indian subcontinent, Asia-Pacific, Eastern Mediterranean, and Northern and Eastern Europe. In Africa, 10-20% prevalence was mostly observed .

The majority of children with asthma have stable disease, and only a minority experience exacerbations needing hospitalization or emergency room visits. In older children, recent advances in treatment seem to have reduced chronic morbidity as well as the number of acute exacerbations. In infants and younger children, this goal may be more difficult to achieve, given the heterogeneity of obstructive lung disease in this age group. Viral wheeze is a very common clinical scenario in young children, and identification and proper treatment of subjects with potential for development of asthma and future exacerbations is still an unresolved challenge. Even if severe asthma exacerbations are relatively common, mortality from asthma in children is rare and declining. In the United Kingdom the mortality rate for children 0-14 years is less than one per 100.000 children per year. In contrast, there has been a vast increase in the economic costs associated with asthma. However, the main economic burden of childhood asthma is linked to indirect costs, long-term follow up and medication, and not to hospitalization .

Acute severe asthma represents one of the most common medical emergency situations and the most serious clinical presentation of asthma. Asthma is typically characterized by the presence of severe respiratory distress due to an asthma episode that requires the use of bronchodilators, oxygen and corticosteroids. Asthma attack can be severe and even life threatening. Features of acute severe attack include; Peak expiratory flow (PEF) 33-50% of best (use % predicted if recent best unknown), tachycardia and tachypnea. Life threatening attack includes pulse oxymetry <92%, Silent chest, cyanosis, or feeble respiratory effort, Arrhythmia or hypotension Exhaustion, altered consciousness. A severe asthma exacerbation can usually be presented clinically with dyspnea at rest; interferes with conversation and peak expiratory flow rate (PEFR) < 40%, usually requires hospitalization .

Acute severe asthma is one of the most common medical emergency situations in childhood, and physicians caring for acutely ill children are regularly faced with this condition. The cornerstones of the management of acute asthma in children are rapid administration of oxygen, inhalations with bronchodilators and systemic corticosteroids. Inhaled bronchodilators may include selective b2-agonists, adrenaline and anticholinergics. Additional treatment in selected cases may involve intravenous administration of theophylline, b2-agonists and magnesium sulphate. Both non-invasive and invasive ventilation may be options when medical treatment fails to prevent respiratory failure. It is important that relevant treatment algorithms exist, applicable to all levels of the treatment chain and reflecting local considerations and circumstances .

Despite recent progress in the treatment of chronic asthma in childhood, acute exacerbations will continue to occur. Physicians working within the field of pediatric emergency medicine will therefore continue to be exposed to this clinical scenario. The cornerstones of acute asthma management in childhood remain rapid onset of oxygen treatment, inhalation of bronchodilators and systemic corticosteroids. Short-acting bronchodilators provide immediate relief of asthma symptoms and effects last four to six hours. The most commonly used short-acting bronchodilator for asthma is albuterol. These medications work quickly, and help to control symptoms of severe asthma attack. The doses as well as the way of delivery are important to reach the best bronchodilator effect. The amount of product that effectively reaches the bronchi is relatively small as 0.1% to 11%, respectively using a lung simulator . Despite this high variation of the amount of product delivery to the patient and the narrow limits of dose between benefice and side effects, the aerosolized route remained the preferred one even in severe cases .

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-16 years.
* Patient with severe asthma (maximum expiratory flow <50%).
* Patient admitted to pediatric emergency.
* Patient who has agreed to participate, as well as the parents or legal guardian.

Exclusion Criteria:

Chronic respiratory failure, infectious disease, heart disease.

* Refusal to participate in the study.
* No affiliation to a social security scheme (beneficiary or beneficiary).
* Immediate intubation criteria

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The main analysis criteria is the Peak expiratory flow (PEF) value performed before the first aerosol of salbutamol aerosols using Jet or Aerogen spray. | 2 minutes
  before the first nebulization
The main analysis criteria is the Peak expiratory flow (PEF) value performed after the first aerosol of salbutamol aerosols using Jet or Aerogen spray. | 2 minutes
  after the first nebulization
The main analysis criteria is the Peak expiratory flow (PEF) value performed after the second aerosol of salbutamol aerosols using Jet or Aerogen spray. | 2 minutes
  after the second nebulization
The main analysis criteria is the Peak expiratory flow (PEF) value performed after the third aerosol of salbutamol aerosols using Jet or Aerogen spray. | 2 minutes
  after the third nebulization

CONTACTS AND LOCATIONS:
Overall Officials: Jean BERGOUNIOUX, MD, Principal Investigator — APHP

IPD SHARING:
Plan to Share IPD: No